CLINICAL TRIAL: NCT05314647
Title: Effects of Lutein Supplementation on Cognition and Vision in Healthy Children With Screen Time Exposure: A Randomized Controlled Trial
Brief Title: Lutein Supplementation in Healthy Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northcentral University (Other)
Responsible Party: Principal Investigator, Brenda Fonseca, Principal Investigator, Northcentral University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NorthcentralU
Record Dates: First submitted 2022-03-05; First posted 2022-04-06 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Eye Fatigue; Diet, Healthy; Cognitive Change
Keywords: lutein; carotenoids; blue light; screen time; digital stress
MeSH Terms: conditions — Asthenopia | interventions — Lutein

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Each participant will be assigned to a group based on a permuted block randomization stratified by participant self-reported sex. Participants may identify male, female or other. If other is selected, assignment as male or female for randomization purposes will be determined by a coin flip. Randomized block lists with a size of 4 will be prepared using a computer generated random number sequence, http://www.jerrydallal.com/random/assigndoc.htm#num (J. Kim & Shin, 2014). Based on group placement, participants will be provided with Bottle A or Bottle B of gummies to last for the next 90 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lutein (Experimental): 5 mg lutein gummy taken daily for 180 days
  Interventions: Dietary Supplement: lutein
- Placebo (Placebo Comparator): 0 mg lutein gummy taken daily for 180 days
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: lutein — daily dose of 5 mg lutein
  Other Names: FloraGLO Lutein
  Arms: Lutein
Dietary Supplement: placebo — daily dose of 0 mg lutein
  Arms: Placebo

SUMMARY:
This is a single site, randomized, double-blind placebo controlled parallel arm study assessing the effects of 6 months lutein supplementation on cognitive and visual outcomes in healthy children exposed to excessive digital screen time.

DETAILED DESCRIPTION:
Studies in humans and primates have also shown that appropriate daily intake of lutein provides protection to the eyes from blue light from screen time devices such as computers, televisions and phones. It has been well-documented that children are spending far over the recommended two hours screen time per day and excessive exposure to the high energy blue light associated with digital devices has been shown to cause both short-term and long-term visual damage as well as disruption to the sleep cycle. With a globally aging population, if this deficit is not addressed adequately early on in life then there will be substantial public health consequences. A recent study predicted that if individuals were to consume the recommended levels of lutein and zeaxanthin daily, there would be a seven percent reduced risk for age related eye disease and a potential savings of over five billion US dollars annually.

ELIGIBILITY:
Inclusion Criteria:

* Age of 8 to 16 years
* guardian-reported general good health
* guardian-reported 4 hours or more of digital screen time daily

Exclusion Criteria:

* Currently using a supplement containing lutein or zeaxanthin

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Macular Pigment Optical Density - heterochromatic flicker photometry | 6 months
  Level of macular carotenoids deposited in the eye measured using the psychophysical technique of heterochromatic flicker photometry (QuantifEye MPS-II Device). Minimum score of 0, no maximum. Average values range from 0.0 to 1.0. Higher numbers represent greater macular pigment.
Macular Pigment Optical Density - haidinger's brushes | 6 months
  Level of macular carotenoids deposited in the eye measured using haidinger's brushes (Azul Optics MP-Eye Device). Minimum score of 0, maximum score of 10. Higher values represent greater macular pigment.

SECONDARY OUTCOMES:
Digital Eye strain change from baseline | 6 months
  Visual Fatigue Scale total score. Minimum score of 6, Maximum score of 24. Higher scores indicate higher levels of digital eye strain.
  Benedetto, S., Drai-Zerbib, V., Pedrotti, M., Tissier, G., & Baccino, T. (2013). E-readers and visual fatigue. PLoS One, 8(12)
Sleep score change from baseline | 6 months
  Total score on the Cleveland Adolescent Sleepiness Questionnaire. Minimum score of 16, Maximum score of 80. Higher scores indicate greater sleepiness.
  Spilsbury, J. C., et al. (2007). "The Cleveland adolescent sleepiness questionnaire: a new measure to assess excessive daytime sleepiness in adolescents." J Clin Sleep Med 3(6): 603-612.
Verbal Fluency | 6 months
  Letter and semantic fluency using letter and animal naming. Total number of words names in a 60 second time frame. Higher score indicates greater verbal fluency

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McNamara, PhD, Study Chair — Northcentral University
Locations (1):
- Kemin Industries, Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: No